CLINICAL TRIAL: NCT00420524
Title: An Open-label, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Patupilone in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Function
Brief Title: A Study of Patupilone in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2121
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2011-12

CONDITIONS: Advanced Malignancies; Tumors
Keywords: EPO; Patupilone; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — epothilone B

ARMS (3):
- Arm A (Normal liver function) (Experimental)
  Interventions: Drug: Patupilone/EPO906
- Arm B (Mild liver dysfunction) (Experimental)
  Interventions: Drug: Patupilone/EPO906
- Arm C (Moderate liver dysfunction) (Experimental)
  Interventions: Drug: Patupilone/EPO906

INTERVENTIONS:
Drug: Patupilone/EPO906

SUMMARY:
This phase I study will determine the pharmacokinetic profile of patupilone in patients with mild or moderately impaired hepatic function within 2 cycles of treatment. The study population for this trial consists of patients with a documented advanced solid tumor. Patients will be stratified into 3 groups: those with normal liver function, and those with mild or moderate liver dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* World Health Organization (WHO) Performance Status score of: 0 - you are fully active and more or less as you were before your illness; 1 - you cannot carry out heavy physical work, but can do anything else; or 2 - you are up and about more than half the day, you can look after yourself, but are not well enough to work.
* Life expectancy of 3 months or more
* Patients with measurable or evaluable disease who have histologically documented advanced solid tumor and who have progressed after systemic therapy or for whom standard systemic therapy does not exist

Exclusion Criteria:

* Severe and/or uncontrolled medical disease
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Presence of any other active or suspected acute or chronic uncontrolled infection
* Severe cardiac insufficiency, with uncontrolled and/or unstable cardiac or coronary artery disease
* History of another malignancy within 5 years prior to study entry, except for curatively treated non-melanotic skin cancer or cervical cancer in situ

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-01; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To assess the effect of hepatic impairment on the pharmacokinetics of patupilone and its metabolite | After completion of the study (approximately 6 weeks from treatment)
To determine the maximum tolerated dose of patupilone in patients with hepatic impairment | After completion of the study (approximately 6 weeks from treatment)

SECONDARY OUTCOMES:
To correlate the level of hepatic dysfunction to observed toxicity and pharmacokinetics | After completion of the study (approximately 6 weeks from treatment)
Safety and tolerability in patients with hepatic impairment will be assessed by adverse events (AEs), serious adverse events (SAEs) and out of range lab values | After completion of the study (approximately 6 weeks from treatment)
To evaluate the preliminary anti-tumor activity which will be assessed by radiological scans every 6 weeks | After completion of the study (approximately 6 weeks from treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (4):
- United States (4):
  - University of California San Diego/Moores Cancer Center, La Jolla, California
  - Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Institute for Drug Development Cancer Therapy & Research Center/The University of Texas Health Science, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- See also: Results can be found for CEPO906A2121 on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4926